CLINICAL TRIAL: NCT02954276
Title: A Randomized, Open Label, Crossover, Bioavailability Study to Compare Omexa Sumatriptan Transmucosal Sublingual Tablet Versus Commercial Imitrex® Sumatriptan Oral Tablet in Healthy Volunteers
Brief Title: Comparative Bioavailability Study of Omexa Sumatriptan vs. Imitrex® in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Targia Pharmaceuticals Ltd. (Industry)
Collaborators: SoluBest Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SB1705; 0189-15-WOMC (Other: Wolfson Medical Center, Holon, Israel)
Record Dates: First submitted 2016-10-31; First posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Migraine
Keywords: safety
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 75 mg Omexa sumatriptan sublingual tablet (Experimental)
  Interventions: Drug: Omexa Sublingual Sumatriptan tablet
- 100 mg Imitrex oral tablet (Active Comparator)
  Interventions: Drug: Imitrex Oral Product

INTERVENTIONS:
Drug: Omexa Sublingual Sumatriptan tablet — 75 mg
  Arms: 75 mg Omexa sumatriptan sublingual tablet
Drug: Imitrex Oral Product — 100 mg
  Other Names: Sumatriptan
  Arms: 100 mg Imitrex oral tablet

SUMMARY:
the trial is a randomized, open label, crossover, single-administration bioavailability study to compare the pharmacokinetic parameters of Omexa sumatriptan transmucosal sublingual tablet versus commercial Imitrex® sumatriptan oral tablet in 14 healthy volunteers.

DETAILED DESCRIPTION:
Volunteers will randomly receive either the commercial oral tablet 100 mg Imitrex® or 75 mg Omexa sublingual tablet under fasted conditions. One week following the first administration, the volunteers will receive the alternative treatment.

Blood samples will be collected at each visit before drug administration and at 5, 15, 30, 45, 60, 90, 120, 240, 360 and 480 min after drug administration, in order to characterize the drug's absorption and pharmacokinetics, as well as to evaluate Omexa formulation safety.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent
2. Man and women volunteers 18-55 years of age
3. Healthy with no clinically relevant abnormalities in the opinion of the investigator as determined by medical history, physical examination, urine analysis and vital signs.
4. Have a BMI of 18-32 kg/m2, inclusive, and a body weight of not less than 50 kg
5. Women of child-bearing potential who agree to use double contraceptive 14 days prior to the study, during whole duration of the study and 30 days after completion of the study.
6. The volunteer agrees to abstain from alcohol intake 48 hours before each administration of study agent and during inpatient portion of the study
7. The volunteer agrees not to consume food or beverages containing, grapefruit or grapefruit juice 72 hours prior to study treatment and until after the last pharmacokinetic (PK) sample is collected
8. The volunteer agrees to frequent blood withdrawal
9. The volunteer doesn't have history of fear of needles and injections, or hemophobia (fear of blood)

Exclusion Criteria:

1. Pregnant or breast-feeding women (women of child bearing potential must use double contraceptive and have the results of a negative pregnancy test recorded prior to study drug administration)
2. Have a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA)
3. Volunteers with two or more risk factors for ischemic heart disease
4. History of seizures
5. History of moderate to severe hypertension or mild uncontrolled hypertension or systolic blood pressure above 140 or diastolic above 90 during screening visit
6. Currently or history of disease or dysfunction of the pulmonary, cardiovascular, endocrine, hematologic, neurological, immune, gastrointestinal, genitourinary, or other body system that is clinically significant in the opinion of the Investigator.
7. History of hypersensitivity or allergies to any drug compound, including Sumatriptan, any of its components or sulphonamides (Appendix 1).
8. History of traumatic surgery within 12 weeks prior to screening, pre-planned surgery or procedures that would interfere with the conduct of the study.
9. Have an acute illness within 7 days prior to study treatment or have had a major illness or hospitalization within 1 month prior to study treatment.
10. History (within 1 year) of alcohol or drug abuse.
11. Volunteers who are heavy smokers (more than 10 cigarettes a day) or use of nicotine-replacement therapy
12. History of abnormal values for hematology, clinical chemistry, or urine analysis during six months prior to treatment considered clinically significant by the Investigator.
13. Positive test for HIV antibodies at screening
14. Positive HBsAg test at screening, or volunteers that did not bring a certificate for three doses of Hepatitis B vaccination.
15. Known history of positive serology test for hepatitis C virus antibody (anti-HCV)
16. Positive urine drug screen for substances of abuse including cocaine, cannabinoids, amphetamines, benzodiazepines, Subutex (BUP), opiates, and methadone at screening.
17. Have donated blood or experienced significant blood loss (volume > 500 mL) within 3 months prior to screening, or is planning to donate within 2 months after completion of the study.
18. Use of any monoamine oxidase inhibitors (MAOI) within 28 days prior to study treatment .
19. Use of any prescription medications/products, except hormonal contraceptives, within 14 days prior to each of the study treatments.
20. Use of any over the counter (OTC), nonprescription preparation (including minerals and phytotherapeutic/herbal/plant-derived preparations), within 14 days prior to each of the study treatments, with the exception of ibuprofen, and acetaminophen used at recommended doses.
21. Participation in any other investigational study in which receipt of an investigational study treatment occurred within 4 weeks prior to dosing, or plan to participate in an investigational study less than 1 month after completion of the study.
22. Any condition that in the opinion of the Investigator would complicate or compromise the study, or the well-being of the volunteer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time to reach peak plasma concentration (Tmax) | Predose, 5, 15, 30, 45, 60, 90, 120, 240, 360 and 480 min post-dose
Peak Plasma concentration (Cmax) | Predose, 5, 15, 30, 45, 60, 90, 120, 240, 360 and 480 min post-dose
Area under the curve (AUC) | Predose, 5, 15, 30, 45, 60, 90, 120, 240, 360 and 480 min post-dose

SECONDARY OUTCOMES:
Adverse events | Through study completion, an average of 2 months

IPD SHARING:
Plan to Share IPD: No